CLINICAL TRIAL: NCT02813109
Title: Urine Biomarkers for Renal Function Monitoring in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Inha University Hospital (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Juyoung Lee, MD, PhD, Inha University Hospital
Other Study IDs: U-BIO-16
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine

SUMMARY:
The true renal function of preterm infants is difficult to evaluate. Serum creatinine (Cr) levels in infants are unreliable as a detector of renal function in the first few days of life because they may continue to reflect maternal levels. Although few candidates appear to be a useful biomarker for kidney injury, scant reference data on these biomarker in preterm infants exist, and studies have yielded conflicting results. Therefore, we aimed to determine the reliable urinary biomarkers to detect kidney injuries in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* premature infants born before 37 weeks of gestational age

Exclusion Criteria:

* cardiac or renal anomalies
* transferred in 2 days after birth from other hospitals

Ages: 1 Day to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: below gestational age 37 weeks
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
correlation of urinary NGAL (neutrophil-gelatinase-associated lipocalin) with serum creatinine | postnatal 1day
correlation of urinary NGAL (neutrophil-gelatinase-associated lipocalin) with serum creatinine | postnatal 3day
correlation of urinary NGAL (neutrophil-gelatinase-associated lipocalin) with serum creatinine | postnatal 5day
correlation of urinary NGAL (neutrophil-gelatinase-associated lipocalin) with serum creatinine | postnatal 7day

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Inha University Hospital, Incheon
  - Hallym University Medical Center - Kangnam, Seoul